CLINICAL TRIAL: NCT06028893
Title: A Real-World Validation Study of Intermittent Photoplethysmography Based Rhythm Monitoring for Atrial Fibrillation Detection
Brief Title: REal-worLd vAlidaTION of PhotoPlehtysmoGraphy (for Atrial Fibrillation Detection)
Acronym: RELATION PPG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Z-2021058-2
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-08

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Photoplethysmography; Single-lead ECG; Electrocardiogram; Digital Health
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Study group (Experimental): All subjects will perform heart rhythm measurements with both diagnostic tests.
  Interventions: Diagnostic Test: Heart rhythm measurements with FibriCheck®; Diagnostic Test: Heart rhythm measurements with Kardia Mobile®

INTERVENTIONS:
Diagnostic Test: Heart rhythm measurements with FibriCheck® — Measurements are performed twice daily, starting 4 weeks before a pulmonary vein isolation procedure (PVI) and ending 4 weeks after the PVI.
Diagnostic Test: Heart rhythm measurements with Kardia Mobile® — Measurements are performed immediately before and after every FibriCheck® measurement.

SUMMARY:
Mobile health solutions for rhythm monitoring (e.g. atrial fibrillation detection) using photoplethysmography (PPG) technology on a smartphone have been developed. This study validates the performance of a digital health application (FibriCheck®) using PPG technology on a smartphone against a single-lead ECG device (Kardia Mobile®).

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled for an ablation procedure for AF, at least 4 weeks after the inclusion.
* Subject provides informed consent.
* Subject understands and agrees to comply with planned study procedures.
* Subject is able to perform measurements of the heart rhythm using the FibriCheck application at home.

Exclusion Criteria:

* Insufficient cognitive or comprehensive level of Dutch to participate to the trial.
* No access to a smartphone or unable to perform FibriCheck measurements at home.
* Pacemaker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity | Two months
  Proportion of true positives tests with FibriCheck® out of all patients with AF on Kardia Mobile®.
Specificity | Two months
  Proportion of true negative tests with FibriCheck® out of all patients in sinus rhythm on Kardia Mobile®.
Overall accuracy (proportion of correct classifications) | Two months
  Proportion of correct classifications with FibriCheck®. Correct classification is provided by Kardia Mobile®.

SECONDARY OUTCOMES:
Positive predictive value | Two months
  Positive predictive value of FibriCheck® measurements relative to Kardia Mobile®.
Negative predictive value | Two months
  Negative predictive value of FibriCheck® measurements relative to Kardia Mobile®.
Sensitivity by heart rate interval | Two months
  Proportion of true positives tests with FibriCheck® out of all patients with AF on Kardia Mobile®.
Specificity by heart rate interval | Two months
  Proportion of true negative tests with FibriCheck® out of all patients in sinus rhythm on Kardia Mobile®.
Accuracy by heart rate interval | Two months
  Proportion of correct classifications with FibriCheck®. Correct classification is provided by Kardia Mobile®.
Proportion of PPG measurements of insufficient quality for rhythm analysis | Two months
  PPG measurements by FibriCheck®.
Proportion of ECG measurements of insufficient quality for rhythm analysis | Two months
  ECG measurements by Kardia Mobile®.
Proportion of PPG measurements of insufficient quality for rhythm analysis by heart rate interval | Two months
  PPG measurements by FibriCheck®.
Proportion of ECG measurements of insufficient quality for rhythm analysis by heart rate interval | Two months
  ECG measurements by Kardia Mobile®.

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No